CLINICAL TRIAL: NCT00408200
Title: A Randomized Trial to Assess the Utility of Empirical Anti-Arrhythmic Drug Therapy to Prevent Atrial Arrhythmia During the 6 Weeks Following Pulmonary Vein Isolation to Treat Paroxysmal Atrial Fibrillation
Brief Title: A Study of the Effectiveness of Anti-Arrhythmic Medications After Atrial Fibrillation Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 805346HUP
Record Dates: First submitted 2006-12-01; First posted 2006-12-06 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Atrial arrhythmia
MeSH Terms: conditions — Atrial Fibrillation | interventions — Propafenone; Flecainide; Sotalol; dofetilide; Catheter Ablation

ARMS (2):
- AAD:YES (Other): Subjects receive membrane-active anti-arrhythmic medication after ablation. See intervention list below.
  Interventions: Drug: propafenone; flecainide; sotalol; dofetilide; Device: Radiofrequency catheter ablation
- AAD:NO (Other): Subjects do not receive membrane-active anti-arrhythmic medications after ablation.
  Interventions: Device: Radiofrequency catheter ablation

INTERVENTIONS:
Drug: propafenone; flecainide; sotalol; dofetilide — Above drugs prescribed per established guidelines for treatment of AF
  Arms: AAD:YES
Device: Radiofrequency catheter ablation — A special catheter that delivers radiofrequency (heat) energy is advanced into the heart and used to destroy small areas of heart tissue responsible for causing atrial fibrillation. All catheters / devices used in the study are FDA approved for human use and currently being used to perform the AF ablation procedure in the United Sates.

SUMMARY:
The purpose of this study is to examine the overall effectiveness of anti-arrhythmic medicines (to control heart rhythm) prescribed after an ablation procedure for atrial fibrillation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder in the US and it is associated with shortness of breath, palpitations, stroke occurrence and increased mortality. Traditional treatment for AF includes anticoagulation, drugs that slow the heart rate and antiarrhythmic agents. More recently, catheter based treatments to address atrial fibrillation have been developed, which involves using radiofrequency energy to isolate the arrhythmogenic foci localized in the pulmonary veins.

During the first weeks following pulmonary vein isolation (PVI), it is not unusual for patients to experience early recurrences of atrial fibrillation or atrial tachycardia due to irritability from the ablation. While these arrhythmias tend to resolve over time, it is nevertheless standard practice to prescribe antiarrhythmic drugs for the first 2-3 months after the intervention to prevent these early recurrences. However, the efficacy of this practice has never been formally evaluated. In addition, we have identified a small group of patients whose atrial tachycardias have terminated after cessation of antiarrhythmic therapy, suggesting that proarrhythmia from these agents may promote reentrant tachycardias in some patients. We therefore designed a study protocol that will evaluate the usefulness of short term antiarrhythmic drug therapy in order to prevent atrial fibrillation and atrial tachycardia episodes during the first 6 weeks following PVI.

The target population of the study includes all patients with paroxysmal atrial fibrillation referred for PVI. After the ablation procedure, patients will be randomized to receive or not receive antiarrhythmic drugs for a period of 6 weeks. Arrhythmia occurrence during this period will be monitored via twice daily transtelephonic monitoring. Clinical visits including a physical exam and 12 lead ECG recording will be scheduled at 6 weeks. The primary endpoint of the study will be a composite endpoint including 1) atrial arrhythmias persisting > 24 hours or requiring initiation of antiarrhythmic therapy 2) need for cardioversion/hospital admission 3) need for repeat ablation or 4) adverse outcome/intolerance of antiarrhythmic agent requiring drug cessation or change during the 6 week follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients meeting ACC/AHA criteria for paroxysmal atrial fibrillation (episodes typically last no more than 7 days and are self-terminating)
* Eligible for pulmonary vein isolation
* Able to tolerate antiarrhythmic medication

Exclusion Criteria:

* Age <18
* Persistent or permanent atrial fibrillation (episodes last >7 days and require cardioversion)
* Antiarrhythmic treatment for indication other than atrial fibrillation
* Contraindication or intolerance to all antiarrhythmic medications
* Primary physician unwilling to withhold antiarrhythmic drugs for duration of the study
* Failure to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward P. Gerstenfeld, MD, Principal Investigator — University of Pennsylvania Health System - Cardiac Electrophysiology
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Roux JF, Zado E, Callans DJ, Garcia F, Lin D, Marchlinski FE, Bala R, Dixit S, Riley M, Russo AM, Hutchinson MD, Cooper J, Verdino R, Patel V, Joy PS, Gerstenfeld EP. Antiarrhythmics After Ablation of Atrial Fibrillation (5A Study). Circulation. 2009 Sep 22;120(12):1036-40. doi: 10.1161/CIRCULATIONAHA.108.839639. Epub 2009 Sep 8. PMID 19738139
- [Derived] Leong-Sit P, Roux JF, Zado E, Callans DJ, Garcia F, Lin D, Marchlinski FE, Bala R, Dixit S, Riley M, Hutchinson MD, Cooper J, Russo AM, Verdino R, Gerstenfeld EP. Antiarrhythmics after ablation of atrial fibrillation (5A Study): six-month follow-up study. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):11-4. doi: 10.1161/CIRCEP.110.955393. Epub 2010 Nov 13. PMID 21076158

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: 12/06 to 3/08.
Pre-assignment Details: Following consent/enrollment, subject and investigator were blinded to treatment arm until after the ablation procedure. Subjects were later withdrawn if the procedure was not completed, or if a disqualifying medication history or other protocol exclusion was identified.
Groups:
- AAD:NO: Subjects do not receive membrane-active anti-arrhythmic medications after ablation.
  Radiofrequency catheter ablation : A special catheter that delivers radiofrequency (heat) energy is advanced into the heart and used to destroy small areas of heart tissue responsible for causing atrial fibrillation. All catheters / devices used in the study are FDA approved for human use and currently being used to perform the AF ablation procedure in the United Sates.
- AAD:YES: Subjects receive membrane-active anti-arrhythmic medication after ablation. See intervention list below.
  Radiofrequency catheter ablation : A special catheter that delivers radiofrequency (heat) energy is advanced into the heart and used to destroy small areas of heart tissue responsible for causing atrial fibrillation. All catheters / devices used in the study are FDA approved for human use and currently being used to perform the AF ablation procedure in the United Sates.
  propafenone; flecainide; sotalol; dofetilide : Above drugs prescribed per established guidelines for treatment of AF
Period: Overall Study
Arm/Group | AAD:NO | AAD:YES
Started | 57 | 53
Completed | 57 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AAD:NO | AAD:YES | Total
Number analyzed (Participants) | 57 | 53 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 53 | 110
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 41 | 37 | 78
Region of Enrollment [Number; unit: participants]
  United States | 57 | 53 | 110

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint: Atrial Arrhythmias Lasting >24 Hrs or Requiring Antiarrhythmic Drug Therapy; Need for Cardioversion/Repeat Ablation During the Study Period; Adverse Outcome/Intolerance of Antiarrhythmic Agent Requiring Cessation or Change of Drug
Time Frame: 6 weeks
Population: Assuming an incidence of the composite primary end point of 40% in the control group and a 50% reduction in the composite primary end point in the drug treatment group, we calculated that 160 patients would have to be included in the study in order to obtain a power of 80% and with a 2-tailed error of 0.05.
Measure: Number; unit: participants
Arm/Group | AAD:NO | AAD:YES
Number analyzed (Participants) | 57 | 53
participants | 24 | 10

2. Secondary Outcome: Freedom From Atrial Arrhythmia at 6 Months Post Procedure.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | AAD:NO | AAD:YES
Number analyzed (Participants) | 57 | 53
participants | 39 | 35
Statistical Analysis 1: Comparison: AAD:NO vs AAD:YES; Test type: Superiority or Other; p < 0.05, Fisher Exact

ADVERSE EVENTS:
Arm/Group | AAD:NO | AAD:YES
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53
Other Adverse Events (participants affected / at risk) | 0/57 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes